CLINICAL TRIAL: NCT02961036
Title: The Role of Supplementary Material in Journal Articles Surveys of Authors, Reviewers and Readers Questionnaire Trial
Brief Title: The Role of Supplementary Material in Journal Articles QT
Acronym: SupMatQT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ThinkWell (Other)
Collaborators: The BMJ (Other); University of Oxford (Other); Queen's University, Belfast (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: ThinkWell
Record Dates: First submitted 2016-11-05; First posted 2016-11-10 (Estimated); Last update posted 2021-03-22 (Actual); Status verified 2021-03

CONDITIONS: Incentive
Keywords: Surveys and Questionnaires

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (7):
- Group 1 Information (Experimental): Group 1 Information about the prize draw incentive for 100% of an Amazon gift (or currency equivalent) in the invitation letter.
  Interventions: Other: Group 1 information
- Group 2 Information (Active Comparator): Group 2 Information about the prize draw incentive for 75% of an Amazon gift (or currency equivalent) in the invitation letter.
  Interventions: Other: Group 2 information
- Group 3 Information (Active Comparator): Group 3 Information about the prize draw incentive for 50% of an Amazon gift (or currency equivalent) in the invitation letter.
  Interventions: Other: Group 3 information
- Group 4 Information (Active Comparator): Group 4 Information about the prize draw incentive for 25% of an Amazon gift (or currency equivalent) in the invitation letter.
  Interventions: Other: Group 4 information
- Group 5 No Information (Active Comparator): Group 5 No Information incentive for an Amazon gift certificate (or currency equivalent) in the invitation letter.
  Interventions: Other: Group 5 no information
- Group A reminder (Experimental): One survey reminder at 14 days
  Interventions: Other: Group A Reminder
- Group B reminders (Active Comparator): Two survey reminders 14 days and 28 days
  Interventions: Other: Group B Reminders

INTERVENTIONS:
Other: Group 1 information — Group 1 prize draw information for participants to win 100% of an Amazon gift card (or currency equivalent) in invitation letter.
  Arms: Group 1 Information
Other: Group 2 information — Group 2 prize draw information for participants to win 75% of an Amazon gift card (or currency equivalent) in invitation letter.
  Arms: Group 2 Information
Other: Group 3 information — Group 3 prize draw information for participants to win 50% of an Amazon gift card (or currency equivalent) in invitation letter.
  Arms: Group 3 Information
Other: Group 4 information — Group 4 prize draw information for participants to win 25% of an Amazon gift card (or currency equivalent) in invitation letter.
  Arms: Group 4 Information
Other: Group 5 no information — Group 5 no Information for participants to enter a draw to win an Amazon gift card (or currency equivalent) in invitation letter.
  Arms: Group 5 No Information
Other: Group A Reminder — One survey reminder at 14 days
  Arms: Group A reminder
Other: Group B Reminders — Two survey reminders one at 14 days and one at 28 days
  Arms: Group B reminders

SUMMARY:
Questionnaires are frequently used in online research, however recruiting, and completion rates of online participants from a variety of cultures and demographic backgrounds can be challenging. The challenge is greater in an online cohort because there is no way to observe the participant beyond what is contributed online. Poor recruiting and completion can result in underpowered research that may not be representative of the sample population. This can trigger an increase in costs as the recruitment period may have to be extended until sample size is reached. When recruiting and completion rates are inadequate studies may have to be terminated and the answer to the research question can remain unknown.

To mitigate these challenges, incentives may be offered in the form of gift certificate draws. There is uncertainty about whether this strategy is effective in online research and if the value of the incentive alters the outcome. A randomised trial can be used to test the intervention to establish an evidence base.

This study (SupMatQT) proposes to link with a large 20,000 person international cohort study (SupMat) that will test the utility and preferences of journal supplementary materials for reviewers, authors,and readers. The research described here will examine the evidence of effect for offering a prize draw incentive on rates of recruitment, and completion for consented participants. All participants will be entered in the draw. Information about the value of the incentive of a prize draw will differ according to what group a participant is randomized to. The entry in the prize draw will not be conditional on levels of participation or group allocation.

The other question researchers will address is what effect do survey reminders have on outcomes? All non-responders will be sent an initial reminder to complete the survey (Group A) and for those who have still not responded a second reminder will be sent 14 days later (Group B). Outcomes will be compared at three time points: for initial response, following reminder 1(Group A), and following reminder 2 (Group B).

DETAILED DESCRIPTION:
The Role of Supplementary Material in Journal Articles is a research collaboration between the BMJ, University of Oxford, and Queen's University Belfast where the research team aims to explore the usage patterns of supplementary materials for journal articles by authors, peer reviewers, and readers and to compare authors, peer reviewers and readers responses to these materials. The large cohort provides a unique opportunity to conduct methodology research with online participants using a nested cohort study defined as a study within a trial (SWAT). The nested study "The Role of Supplementary Material in Journal Articles Questionnaire Study " will explore the effects of recruitment and survey completion when a prize draw for participants is included in the invitation letter.

Large research populations can struggle to recruit participants and to obtain complete data. This can have a direct effect on the robustness of the findings and can undermine the often substantial investment, participants, researchers, and sponsors have made in the research. This research waste may undermine public trust and community enthusiasm for the research process. It may seem logical to offer a prize-winning draw as an incentive but only a trial can give objective information about how well this intervention works. It is cost effective to embed this research at the beginning of an existing large cohort study as funding may not be available to test the intervention as a stand alone question. The additional question of interest addressed will be asking whether one survey reminder or two is more effective in terms of recruitment and survey completion rates. The question is practical as ineffective reminders use researcher resources, increase the burden of participation on the participant and could build resentment if the respondent feels "spammed" whereas the ideal balance of reminders will result in increased recruitment and survey completion rates.

Participants in this cohort are drawn from a convenience sample of BMJ Publishing Group's journals that have a spread of Impact Factors, including the BMJ. Included journals have a website and publish supplementary material.

Devoting time and resources to understand what strategies will mobilize participants to remain motivated to join a study and complete the conditions is good planning and contributes to robust methods that other researchers can replicate. To the investigators' knowledge, no similar work has been conducted solely within the online population of readers, peer reviewers and authors of an academic journal group.

The aims of the study are to test the effect of:

1. Being told you will be entered into a prize draw versus not being told on survey recruitment and completion rates across three surveys (authors, readers, reviewers)
2. Entering participants into a prize draw with different values of monetary incentives on survey recruitment and completion rates across three surveys (authors, readers, reviewers)
3. Sending two survey reminders to each of these incentive groups on survey recruitment and completion rates across three surveys (authors, readers, reviewers)

The research question(s) this research explores is, what effect does the knowledge of being entered into a prize draw have on the rates of recruitment and completion in the study and does varying the value of the incentive influence the outcomes. The study will describe how or if these rates differ between authors, reviewers, and readers. The second question is how does one v two reminders influence recruitment and completion rates.

Participants (authors, reviewers ,and readers) will be invited to take part in the study and will be randomized into one of five trial arms:

All potential participants who are non-responders will receive one reminder to complete the survey (Group A), For those who are still non-responders the initial reminder will be followed by an additional reminder 14 days later (Group B)

Group one will receive information within the invitation letter that they will be entered into a prize draw to win a 100% of an Amazon gift certificate or the currency equivalent.

Group two will receive information within the invitation letter that they will be entered into a prize draw to win a 75% of an Amazon gift certificate or the currency equivalent.

Group three will receive information within the invitation letter that they will be entered into a prize draw to win a 50% of an Amazon gift certificate or the currency equivalent.

Group four will receive information within the invitation letter that they will be entered into a prize draw to win a 25% of an Amazon gift certificate or the currency equivalent.

Group five will not receive any information about the prize draw for an Amazon gift certificate in the invitation letter.

ELIGIBILITY:
Inclusion Criteria:

* Part of SupMat Research
* Corresponding authors of BMJ Group full-length original research submissions in 2013
* BMJ Group Reviewers who completed a review of a manuscript for "original research", "research" or "paper" in 2014.
* BMJ authors, reviewers, and reviewers with a viable email address

Exclusion Criteria:

* Not Part of SupMat Research
* Potential participants who have opted out of BMJ communications
* Participants in BMJ surveys within the last 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2872 (Actual)
Dates: Start 2016-11-15 (Actual); Primary Completion 2017-02-15 (Actual); Study Completion 2019-02-25 (Actual)

PRIMARY OUTCOMES:
Completion | Duration of study up to 60 days
  proportion of questions completed in the questionnaire

SECONDARY OUTCOMES:
Recruitment | Duration of study up to 60 days
  proportion of sample recruited
  • Secondary Outcome Measure: proportion of sample recruited Comparison of recruitment numbers between Groups one through five and Groups A and B

CONTACTS AND LOCATIONS:
Overall Officials: Mike Clarke, PhD, Principal Investigator — Queens University Belfast
Locations (1):
- ThinkWell, Oxford, Oxfordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Data will be shared in aggregated form upon request in order to comply with data protection policies

REFERENCES:
- [Background] Asch DA, Jedrziewski MK, Christakis NA. Response rates to mail surveys published in medical journals. J Clin Epidemiol. 1997 Oct;50(10):1129-36. doi: 10.1016/s0895-4356(97)00126-1. PMID 9368521
- [Background] Kenyon J, Sprague N, Flathers E. The Journal Article as a Means to Share Data: a Content Analysis of Supplementary Materials from Two Disciplines. J Librarianship Scholarly Community 2016;4:eP2112. doi:10.7710/2162-3309.2112
- [Background] Baruch Y, Holtom BC. Survey response rate levels and trends in organizational research. Hum Relations 2008;61:1139-60. doi:10.1177/0018726708094863
- [Background] Cobanoglu C. The effect of incentives in web surveys : application and ethical considerations. Int J Mark Res 2003;45:475-88.
- [Background] Beebe L. Supplemental materials for journal articles: NISO/NFAIS working group. Information Standards Quarterly 2010;22:33-7. doi:10 .3789/isqv22n3.2010.07
- [Background] Education section - Studies Within A Trial (SWAT). J Evid Based Med. 2012 Feb;5(1):44-5. doi: 10.1111/j.1756-5391.2012.01169.x. No abstract available. PMID 23528122
- [Result] Price A, Schroter S, Clarke M, McAneney H. Role of supplementary material in biomedical journal articles: surveys of authors, reviewers and readers. BMJ Open. 2018 Sep 24;8(9):e021753. doi: 10.1136/bmjopen-2018-021753. PMID 30249629